CLINICAL TRIAL: NCT01941082
Title: A Multiple-Center, Non-Randomized, Open-Label, Single- and Multiple-Ascending-Dose, Parallel Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO6867461 Following Intravitreal Administration in Patients With Wet Age-Related Macular Degeneration
Brief Title: A Study of RO6867461 Administered in Single- and Multiple-Ascending Doses in Patients With Wet Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP28936; 2013-001972-40 (EudraCT Number)
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

ARMS (2):
- Part A: RO6867461 (Experimental): Single doses
  Interventions: Drug: RO6867461
- Part B: RO6867461 (Experimental): Multiple doses
  Interventions: Drug: RO6867461

INTERVENTIONS:
Drug: RO6867461 — Single or multiple ascending dose by intravitreal injection

SUMMARY:
This multicenter, non-randomized, open-label, single- and multiple-ascending-dose study will investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of RO6867461 in patients with wet age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 50 years of age
* Patients with age-related macular degeneration (AMD)
* Best corrected visual acuity (BCVA) of 20/40 to 20/400 (Snellen equivalent, on ETDRA charts) inclusive
* Evidence of leakage due to choroidal neovascularization (CNV)

Exclusion Criteria:

* Choroidal neovascularization (CNV) in either eye due to causes other than age related macular degeneration, such as ocular histoplasmosis, trauma, or pathologic myopia
* Known hypersensitivity to ranibizumab, fluorescein, indocyanin green (ICG) or any of the ingredients of the formulation used, or any of the medications used
* Any other restriction according to the use of ranibizumab
* Active intraocular inflammation (grade trace or above) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Ocular safety, assessed by BCVA (EDTRS chart), slitlamp examination, ophthalmoscopy, IOP, fundus photography, SD-OCT, angiography | Part A, 12 weeks; Part B, 20 weeks
Safety: Incidence of adverse events | Part A, 12 weeks; Part B, 20 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration time curve (AUC) | Part A, 12 weeks; Part B, 20 weeks
Pharmacokinetics: Maximum plasma concentration (Cmax) | Part A, 12 weeks; Part B, 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (5):
  - Colorado Springs, Colorado
  - Baltimore, Maryland
  - Dallas, Texas
  - Houston, Texas
  - Charlottesville, Virginia
- United Kingdom (3):
  - Belfast
  - Bristol
  - London